CLINICAL TRIAL: NCT04694352
Title: Effects of Trampoline Exercises Children With Developmental Coordination Disorder
Brief Title: Trampoline Exercises Children With Developmental Coordination Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC00662 Maryam Suleman
Record Dates: First submitted 2020-12-02; First posted 2021-01-05 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2021-01

CONDITIONS: Developmental Coordination Disorder
Keywords: Balance; Developmental coordination disorder; Motor Activity; Quality of Life
MeSH Terms: conditions — Motor Skills Disorders; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Jumping Exercises (Experimental): Jumping in place Jump and clap Jump and reach Jump and twist Jump and turn Half jumping jack Jumping side to side
  Interventions: Other: Jumping Exercises
- Conventional (Active Comparator): Drop and catch a ball Squeeze ball between legs, jump up and catch the ball Walking on a straight line Stand on one leg try to pick object from floor without using hands (do this on both legs) Drop the ball and catch it with both hands Jump up stair with both limbs off the floor simultaneously while holding railing.
  Skipping.
  Interventions: Other: Conventional Physical therapy

INTERVENTIONS:
Other: Jumping Exercises — Jumping in place Jump and clap Jump and reach Jump and twist Jump and turn Half jumping jack Jumping side to side Each exercise done for 1 minute, 5 repetitions is session of 1 hour 15minutes
  Arms: Jumping Exercises
Other: Conventional Physical therapy — Drop and catch a ball Squeeze ball between legs, jump up and catch the ball Walking on a straight line Stand on one leg try to pick object from floor without using hands (do this on both legs) Drop the ball and catch it with both hands Jump up stair with both limbs off the floor simultaneously while holding railing.
  Skipping. At least 5 repetitions for each exercise in session of total 1 hour
  Arms: Conventional

SUMMARY:
RCT in which 28 children with developmental coordination disorder (DCD) were enrolled and equally distributed into two groups; Participants in control group were treated with conventional physical therapy while experimental were given conventional physical therapy in addition to trampoline exercises. Assessment was at 0, 4 and 8 week using developmental coordination disorder questionnaire (DCDQ), pediatric balance scale (PBS) and peads quality of life (PQL)

ELIGIBILITY:
Inclusion Criteria:

* Children with DCD indicated using DCDQ.

Exclusion Criteria:

* No developmental coordination disorder
* declined to participate
* Progressive unstable health condition.

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 28 (Actual)
Dates: Start 2020-08-30 (Actual); Primary Completion 2020-11-28 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
Developmental coordination disorder questionnaire (DCDQ) | 8 weeks
  Developmental Coordination Questionnaire (DCDQ) is a scale to diagnose 5 to 15 year children with DCD and measure their developmental features but through parents reporting, Parents are asked to compare functional task and motor activity of their children with other children
Pediatric balance scale (PBS) | 8 weeks
  Pediatric Balance Scale (PBS) is a scale used to assess child's balance. It is fourteen item scale same as Berg Balance scale.
Peads quality of life (PQL) | 8 weeks
  The Peads quality of life (PQL) Measurement Model is scale for measuring health related quality of life (HRQOL) in children. It has excellent reliability of 0.88 and found measure quality of life in children ranging from healthy to chronic health conditions

CONTACTS AND LOCATIONS:
Overall Officials: Mirza Obaid Baig, Principal Investigator — Riphah International University
Locations (1):
- Federal Government Polyclinic Hospital, Islamabad, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mitsiou M, Giagazoglou P, Sidiropoulou M, Kotsikas G, Tsimaras V, Fotiadou E. Static balance ability in children with developmental coordination disorder. European Journal of Physical Education and Sport. 2016;11:17-23.
- [Background] de Oliveira IS, da Silva Oliveira D, de Azevedo Guendler J, Rocha BM, Sarinho SW. Effectiveness of motor intervention on children with Developmental Coordination Disorder (DCD): A systematic review. Journal of Physical Education and Sport Management. 2017;8(3):32-40.